CLINICAL TRIAL: NCT01627600
Title: The Atahualpa Project, a 3-phase Epidemiologic Survey
Brief Title: Door-to-door Survey of Cardiovascular Health, Stroke and Ischemic Heart Disease in Atahualpa
Acronym: TAP
Status: Completed | Type: Observational
Sponsor: Hospital Clínica Kennedy (Other)
Collaborators: Universidad de Especialidades Espiritu Santo (Other)
Responsible Party: Principal Investigator, Oscar H. Del Brutto, MD, Staff Member, Department of Neurological Sciences, Hospital Clínica Kennedy
Other Study IDs: TAP-001-2012
Record Dates: First submitted 2012-06-15; First posted 2012-06-26 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Stroke; Ischemic Heart Disease
Keywords: stroke; myocardial infarction; cardiovascular health; population study
MeSH Terms: conditions — Stroke; Myocardial Ischemia; Myocardial Infarction

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Atahualpa residents aged ≥ 40 years: All Atahualpa residentes aged 40 ≥ years will be screened by field questionnaires. Then, those with suspected stroke or ischemic heart disease will be evaluated by neurologists and cardiologists. Cardiovascular health metrics will be evaluated in those negative for stroke or ischemic heart disease.

SUMMARY:
The aim of the Atahualpa project is to evaluate the cardiovascular (CVH) status of the inhabitants of a rural village of coastal Ecuador as well as to determine the prevalence and retrospective incidence of stroke and ischemic heart disease. The protocol may be used as a pilot for large-scale studies attempting to evaluate the CVH of rural or even urban centers of Latin America, to implement cost-effective strategies directed to reduce the burden of stroke and cardiovascular diseases in the population at large.

DETAILED DESCRIPTION:
This is a 3-phase epidemiological study. During Phase I, two general physicians and a nurse will perform a door-to-door survey of all Atahualpa residents aged ≥ 40 years. These persons will be eligible for being screened with standardized questionnaires to identify those with suspected stroke or ischemic heart disease, and to evaluate their cardiovascular health (CVH). Persons will be directly interviewed unless aphasic or mentally impaired; in such cases, relatives or caregivers will answer the questions. We plan to use the epidemiologic method of capture-recapture to enhance the detection of all possible cases of stroke and ischemic heart disease [13]. So, besides the door-to-door survey, we will review the medical records from the only one health center of Atahualpa, as well as the original files of our survey performed in 2003 at the same village [12].

In Phase II, certified neurologists and cardiologists will move to Atahualpa to examine all individuals who screened as suspected cases of stroke or ischemic heart disease. In addition, a random sample of 2% of individuals who were considered negative during the screening phase (matched by age and gender to suspected cases) will also undergo a complete neurologic and cardiologic examination to assess possible false negative cases during the survey. In Phase III, all patients with a clinical diagnosis of stroke and ischemic heart disease will be invited to undergo further examination in Guayaquil.

ELIGIBILITY:
Inclusion Criteria:

* Atahualpa residents aged ≥ 40 years

Exclusion Criteria:

* Patients who do not sign the informed consent form

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CVH status will be evaluated in all Atahualpa residents aged ≥ 40 years who did not have history of stroke or ischemic heart disease.
  Certified neurologists and cardiologists will evaluate all individuals who screened as suspected cases of stroke and ischemic heart disease during Phase I of the study, as well as a 2% sample of age- and gender-matched negative individuals.
  All patients with diagnosis of stroke and ischemic heart disease will be invited to undergo complementary exams to achieve more specific diagnosis.
Sampling Method: Probability Sample
Enrollment: 642 (Actual)
Dates: Start 2012-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of cardiovascular health status in Atahualpa residents aged 40 years or more | September 2012 (up to 3 months)
  population will be screened with field questionnaries (3 months), then cardiologists and neurologists will review suspected cases (1 week), then, consented patients will undergo complementary exams

CONTACTS AND LOCATIONS:
Overall Officials: Oscar H Del Brutto, MD, Principal Investigator — Hospital Clinica Kennedy
Locations (2):
- Ecuador (2):
  - Door-to-door survey, Atahualpa, Santa Elena
  - Door-to-Door, Atahualpa, Santa Elena

REFERENCES:
- [Background] Del Brutto OH, Idrovo L, Santibanez R, Diaz-Calderon E, Mosquera A, Cuesta F, Navas C. Door-to-door survey of major neurological diseases in rural Ecuador--the Atahualpa Project: methodological aspects. Neuroepidemiology. 2004 Nov-Dec;23(6):310-6. doi: 10.1159/000080098. Epub 2004 Aug 5. PMID 15297799
- [Background] Del Brutto OH, Idrovo L, Mosquera A, Navas C, Santibanez R, Cuesta F, Diaz-Calderon E. Stroke in rural Ecuador: a three-phase, door-to-door survey. Neurology. 2004 Nov 23;63(10):1974-5. doi: 10.1212/01.wnl.0000145293.04832.78. PMID 15557530
- [Derived] Del Brutto OH, Mera RM, Rumbea DA, Castillo PR. Periodic limb movements in sleep are associated with hippocampal atrophy in stroke-free community-dwelling older adults. Sleep. 2023 Jun 13;46(6):zsad088. doi: 10.1093/sleep/zsad088. No abstract available. PMID 36995971
- [Derived] Del Brutto OH, Mera RM, Costa AF, Rumbea DA, Recalde BY, Castillo PR. Long coronavirus disease-related persistent poor sleep quality and progression of enlarged perivascular spaces. A longitudinal study. Sleep. 2022 Sep 8;45(9):zsac168. doi: 10.1093/sleep/zsac168. No abstract available. PMID 35878737
- [Derived] Del Brutto OH, Mera RM, Costa AF, Recalde BY, Castillo PR. Sleep quality deterioration in middle-aged and older adults living in a rural Ecuadorian village severely struck by the SARS-CoV-2 pandemic. A population-based longitudinal prospective study. Sleep. 2021 Aug 13;44(8):zsab041. doi: 10.1093/sleep/zsab041. PMID 33608714
- [Derived] Del Brutto OH, Mera RM, Penaherrera E, Costa AF, Penaherrera R, Castillo PR. On the Association Between Sleep Quality and Arterial Stiffness: A Population Study in Community-Dwelling Older Adults Living in Rural Ecuador (The Atahualpa Project). J Clin Sleep Med. 2019 Aug 15;15(8):1101-1106. doi: 10.5664/jcsm.7798. PMID 31482831
- [Derived] Del Brutto OH, Castillo PR, Sedler MJ, Del Brutto VJ, Zambrano M, Mera RM, Wright CB, Rundek T. Reasons for Declining Consent in a Population-Based Cohort Study Conducted in a Rural South American Community. J Environ Public Health. 2018 Nov 26;2018:8267948. doi: 10.1155/2018/8267948. eCollection 2018. PMID 30598669